CLINICAL TRIAL: NCT03432143
Title: Community Members as Reviewers of Medical Journal Manuscripts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Ash Sehgal, Investigator, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB17-00374
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Peer Review, Research
Keywords: Peer Review; Community-Based Research; Community Perspectives

STUDY DESIGN:
Intervention Model Description: 24 community members will receive training and mentoring in reviewing manuscripts. The trial will involve 568 manuscripts that will be randomly assigned to two groups using a random number generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Reviewers (Experimental): 24 community members will receive training and mentoring in reviewing manuscripts. Approximately 284 manuscripts will be randomized into the intervention group over the duration of the study. Manuscripts will be reviewed by both a community member and scientific reviewers.
  Interventions: Other: Community Reviewers
- Scientific Reviewers Only (No Intervention): Approximately 284 manuscripts will be randomized into the control group over the duration of the study. Manuscripts will be reviewed by multiple scientific reviewers. Community reviewers will not be involved in reviewing these manuscripts.

INTERVENTIONS:
Other: Community Reviewers — Intervention manuscripts will be reviewed by both a trained community member and scientific reviewers. Community reviewers will follow each journal's instructions regarding electronic access to manuscripts, use of drop-down menus and free-text boxes to address specific aspects of the review, and completion within the time frame specified by the journal.The journal editorial team will use all reviews to make decisions about acceptance, revision, or rejection of manuscripts.
  Arms: Community Reviewers

SUMMARY:
Manuscripts submitted to medical journals are typically reviewed by physicians or researchers, with no input from patients or other community members. However, involvement of community members in other phases of the research process suggests that they provide distinct and useful expertise. Such involvement may lead to enhanced understanding of community priorities, refinement of study designs to minimize participant burden, and increased recruitment and retention of subjects.

The investigators propose a randomized controlled trial involving 24 community members who will receive training and mentoring in reviewing manuscripts. A total of 568 manuscripts submitted to 2 medical journals will be randomly assigned to an intervention or control group. Intervention manuscripts will be reviewed by both a community member and by scientific reviewers while control manuscripts will be reviewed only by scientific reviewers. Journal editorial teams will use all reviews to help them make decisions about acceptance, revision, or rejection of manuscripts.

DETAILED DESCRIPTION:
Manuscripts submitted to medical journals are typically reviewed by physicians or researchers, with no input from patients or other community members. However, involvement of community members in other phases of the research process suggests that they provide distinct and useful expertise. Such involvement may lead to enhanced understanding of community priorities, refinement of study designs to minimize participant burden, and increased recruitment and retention of subjects. In general, community involvement in research is more common in the earlier phases of the research process (selection of research question and development of a study protocol) and less common in later phases (dissemination and implementation of findings). In the investigators' previous work, they conducted a pilot study that recruited and trained community members to review medical journal manuscripts. They found that community reviewers were much more likely than scientific reviewers to comment on i) the relevance of the study to patients and communities, ii) the diversity and complexity of the study participants, iii) the social context of the condition studied, and iv) barriers to implementation of study findings by patients and communities.

The investigators now propose a randomized controlled trial involving 24 community members who will receive training and mentoring in reviewing manuscripts. A total of 568 manuscripts submitted to 2 medical journals will be randomly assigned to an intervention or control group. Intervention manuscripts will be reviewed by both a community member and by scientific reviewers while control manuscripts will be reviewed only by scientific reviewers. Community reviewers will follow each journal's instructions regarding electronic access to manuscripts, use of drop-down menus and free-text boxes to address specific aspects of the review, and completion within the time frame specified by the journal. Journal editorial teams will use all reviews to help them make decisions about acceptance, revision, or rejection of manuscripts. Quantitative and qualitative analyses will i) compare the content of community and scientific reviews, ii) determine the usefulness of community reviews to journal editors, and iii) explore how community reviewer comments are integrated into published articles.

The proposed project is a novel approach to engaging health disparity populations and other community members in dissemination of research findings. This approach has the potential to provide new and distinct perspectives, to increase the quality and relevance of articles published in medical journals, and to enhance dissemination and implementation of research findings.

Primary Aim A. To compare community member reviews with those of scientific reviewers.

Hypothesis: Compared to scientific reviewers, community reviewers will be more likely to comment on relevance to patients and communities, subject diversity, social context, and implementation barriers.

Primary Aim B. To determine the usefulness of community member reviews to editors.

Hypothesis: Editors will report utilizing community reviewer comments in manuscript decisions.

Secondary Aim C. To explore how community reviews are integrated into published articles.

Hypothesis: Community perspectives that were not present in manuscripts at the time of original submission will subsequently be discernible in published articles.

ELIGIBILITY:
Community Reviewer Eligibility:

Inclusion Criteria:

* 18 years or older
* At least a high school diploma
* Proficient in English speaking, reading, and writing
* Computer access
* Personal experience (having the condition or being a caregiver to someone with the condition) with 1 or more of these conditions: Cancer, diabetes, dementia, heart disease, hypertension, liver disease, lung disease, kidney disease, and stroke

Exclusion Criteria:

* Children under 18 years of age
* Non-high school graduates
* Individuals who work in health care settings
* Individuals who have formal training in health care or scientific research

Manuscript Eligibility:

Inclusion Criteria:

* Full length
* Original research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
To compare community member reviews with those of scientific reviewers. | 5 years
  The investigators will examine community and scientific reviewer ratings of intervention group manuscripts, including overall recommendations and ratings of specific aspects of the manuscripts. The overall recommendation categories will be converted into a 4 point Likert scale and combine data across journals.

SECONDARY OUTCOMES:
To determine the usefulness of community member reviews to editors. | 5 years
  The investigators will examine editor ratings of the usefulness of intervention group manuscript reviews submitted by community and scientific reviewers. The investigators will use qualitative analyses to identify specific themes present in editors' responses to open-ended questions about the usefulness of community reviews.

OTHER OUTCOMES:
To explore how community reviews are integrated into published articles. | 5 years
  The investigators will examine how specific community reviewer comments are addressed by authors. They will also examine how often community and patient perspectives are present in published articles.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini Sehgal, Principal Investigator — Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Israel BA, Schulz AJ, Parker EA, Becker AB. Review of community-based research: assessing partnership approaches to improve public health. Annu Rev Public Health. 1998;19:173-202. doi: 10.1146/annurev.publhealth.19.1.173. PMID 9611617
- [Background] Minkler M. Community-based research partnerships: challenges and opportunities. J Urban Health. 2005 Jun;82(2 Suppl 2):ii3-12. doi: 10.1093/jurban/jti034. Epub 2005 May 11. PMID 15888635
- [Background] Caron-Flinterman JF, Broerse JE, Teerling J, Bunders JF. Patients' priorities concerning health research: the case of asthma and COPD research in the Netherlands. Health Expect. 2005 Sep;8(3):253-63. doi: 10.1111/j.1369-7625.2005.00337.x. PMID 16098155
- [Background] Hewlett S, Wit Md, Richards P, Quest E, Hughes R, Heiberg T, Kirwan J. Patients and professionals as research partners: challenges, practicalities, and benefits. Arthritis Rheum. 2006 Aug 15;55(4):676-80. doi: 10.1002/art.22091. No abstract available. PMID 16874772
- [Background] Resnik DB, Kennedy CE. Balancing scientific and community interests in community-based participatory research. Account Res. 2010 Jul;17(4):198-210. doi: 10.1080/08989621.2010.493095. PMID 20597018
- [Background] Wallerstein NB, Duran B. Using community-based participatory research to address health disparities. Health Promot Pract. 2006 Jul;7(3):312-23. doi: 10.1177/1524839906289376. Epub 2006 Jun 7. PMID 16760238
- [Background] Fleurence RL, Forsythe LP, Lauer M, Rotter J, Ioannidis JP, Beal A, Frank L, Selby JV. Engaging patients and stakeholders in research proposal review: the patient-centered outcomes research institute. Ann Intern Med. 2014 Jul 15;161(2):122-30. doi: 10.7326/M13-2412. PMID 25023251
- [Background] Domecq JP, Prutsky G, Elraiyah T, Wang Z, Nabhan M, Shippee N, Brito JP, Boehmer K, Hasan R, Firwana B, Erwin P, Eton D, Sloan J, Montori V, Asi N, Dabrh AM, Murad MH. Patient engagement in research: a systematic review. BMC Health Serv Res. 2014 Feb 26;14:89. doi: 10.1186/1472-6963-14-89. PMID 24568690
- [Background] Forsythe LP, Frank L, Walker KO, Anise A, Wegener N, Weisman H, Hunt G, Beal A. Patient and clinician views on comparative effectiveness research and engagement in research. J Comp Eff Res. 2015 Jan;4(1):11-25. doi: 10.2217/cer.14.52. PMID 25565066
- [Background] Reich SM, Reich JA. Cultural competence in interdisciplinary collaborations: a method for respecting diversity in research partnerships. Am J Community Psychol. 2006 Sep;38(1-2):51-62. doi: 10.1007/s10464-006-9064-1. PMID 16807789
- [Background] Supple D, Roberts A, Hudson V, Masefield S, Fitch N, Rahmen M, Flood B, de Boer W, Powell P, Wagers S; U-BIOPRED PIP group. From tokenism to meaningful engagement: best practices in patient involvement in an EU project. Res Involv Engagem. 2015 Jun 25;1:5. doi: 10.1186/s40900-015-0004-9. eCollection 2015. PMID 29062494
- [Background] Barber R, Boote JD, Parry GD, Cooper CL, Yeeles P, Cook S. Can the impact of public involvement on research be evaluated? A mixed methods study. Health Expect. 2012 Sep;15(3):229-41. doi: 10.1111/j.1369-7625.2010.00660.x. Epub 2011 Feb 17. PMID 21324054
- [Background] Staley K. 'Is it worth doing?' Measuring the impact of patient and public involvement in research. Res Involv Engagem. 2015 Jul 31;1:6. doi: 10.1186/s40900-015-0008-5. eCollection 2015. PMID 29062495
- [Background] Wright D, Foster C, Amir Z, Elliott J, Wilson R. Critical appraisal guidelines for assessing the quality and impact of user involvement in research. Health Expect. 2010 Dec;13(4):359-68. doi: 10.1111/j.1369-7625.2010.00607.x. PMID 20629767
- [Background] Frank L, Forsythe L, Ellis L, Schrandt S, Sheridan S, Gerson J, Konopka K, Daugherty S. Conceptual and practical foundations of patient engagement in research at the patient-centered outcomes research institute. Qual Life Res. 2015 May;24(5):1033-41. doi: 10.1007/s11136-014-0893-3. Epub 2015 Jan 6. PMID 25560774
- [Derived] Huml AM, Albert JM, Beltran JM, Berg KA, Collins CC, Hood EN, Nelson LC, Perzynski AT, Stange KC, Sehgal AR. Community Members as Reviewers of Medical Journal Manuscripts: a Randomized Controlled Trial. J Gen Intern Med. 2023 May;38(6):1393-1401. doi: 10.1007/s11606-022-07802-z. Epub 2022 Sep 26. PMID 36163530